CLINICAL TRIAL: NCT05595278
Title: Detrmination of the Relationship Between Red Cell Distribution Width ,NT-proBNP and cTnT in Acute Myocardial Infraction Patients
Brief Title: Red Cell Distribution Width,,NT-proBNP and cTnT in Acute Myocardial Infraction Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hemat Kamel Maarouf, Resident doctor at clinical and chemical pathology department, Sohag University
Other Study IDs: Soh-Med-2210-05
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: (CBC) ,(NT-proBNP) ,(cTnT) — complete blood count (CBC) including RDW with N-terminal pro-B-type natriuretic peptide (NT-proBNP) and cardiac troponin T (cTnT) in a cohort of acute myocardial infarction (AMI) patients.

SUMMARY:
the study is to investigate the relationship of several parameters of complete blood count (CBC) including RDW with N-terminal pro-B-type natriuretic peptide (NT-proBNP) and cardiac troponin T (cTnT) in a cohort of acute myocardial infarction (AMI) patients.

DETAILED DESCRIPTION:
Patients and methods:

* Type of study: Observational prospective study
* Place of study: Sohag cardiology and gastroenterology center, department of cardiology and cardiac care unit.
* Ethical considerations: This research will be revised by the Scientific Ethical Committee of Sohag University Hospital. Consents will be taken from all patients.
* Study Methods:

  * A prospective study on 30 patients diagnosed as acute myocardial infarction on which measurement of CBC, serum NT-proBNP, and cTnT levels will be performed at the time of admission and by the time of discharge.
  * All patients included in the study will be subjected to:

    1. Full history:

       1. Personal history: e.g. age, sex and smoking.
       2. Family history of cardiac diseases
       3. Medical history of: Hypertension, Ischemic heart disease, prior coronary artery bypass grafting, Prior Percutaneous coronary intervention, Prior Stroke, Prior Atrial fibrillation, therapeutic history
    2. Detailed clinical examination
    3. Electrocardiogram
    4. Laboratory investigation:

       1. Routine investigation in the form of CBC including RDW
       2. Specific investigation which include NT-proBNP and cTnT

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as acute myocardial infarction and admitted to department of cardiology and cardiac care unit at Sohag cardiology and gastroenterology center according to inclusion and exclution criteria

Exclusion Criteria:

Patient with:

* Decompensated heart failure
* Pulmonary hypertention
* Acute pulmonary embolism
* Septic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • All patients included in the study will be subjected to:
  1. Full history:
     1. Personal history: e.g. age, sex and smoking.
     2. Family history of cardiac diseases
     3. Medical history of: Hypertension, Ischemic heart disease, prior coronary artery bypass grafting, Prior Percutaneous coronary intervention, Prior Stroke, Prior Atrial fibrillation, therapeutic history
  2. Detailed clinical examination
  3. Electrocardiogram
  4. Laboratory investigation:
     1. Routine investigation in the form of CBC including RDW
     2. Specific investigation which include NT-proBNP and cTnT
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-13 (Estimated); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-07-13 (Estimated)

PRIMARY OUTCOMES:
(CBC) | 6 months
  measurement of CBC will be performed at the time of admission and by the time of discharge.
(NT-proBNP | 6 months
  measurement of serum NT-proBNP levels will be performed at the time of admission and by the time of discharge.
(cTnT) | 6 months
  measurement of cTnT levels will be performed at the time of admission and by the time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nascimento BR, Brant LCC, Marino BCA, Passaglia LG, Ribeiro ALP. Implementing myocardial infarction systems of care in low/middle-income countries. Heart. 2019 Jan;105(1):20-26. doi: 10.1136/heartjnl-2018-313398. Epub 2018 Sep 29. PMID 30269080
- [Background] Barberi C, van den Hondel KE. The use of cardiac troponin T (cTnT) in the postmortem diagnosis of acute myocardial infarction and sudden cardiac death: A systematic review. Forensic Sci Int. 2018 Nov;292:27-38. doi: 10.1016/j.forsciint.2018.09.002. Epub 2018 Sep 17. PMID 30269044
- [Background] Alaour B, Liew F, Kaier TE. Cardiac Troponin - diagnostic problems and impact on cardiovascular disease. Ann Med. 2018 Dec;50(8):655-665. doi: 10.1080/07853890.2018.1530450. Epub 2018 Nov 21. PMID 30265127